CLINICAL TRIAL: NCT03649867
Title: What Have Been the Experiences of Female Survivors of Interpersonal Trauma on the Survive & Thrive Course
Acronym: EoFSoITotS&TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Dr Lucie Bartoskova, Counselling Psychologist, NHS Tayside
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3-003-18
Record Dates: First submitted 2018-08-20; First posted 2018-08-28 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Interpersonal Trauma

STUDY DESIGN:
Intervention Model Description: Qualitative Study - semi-structured interviews
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi-structured interview (Other): Each female patient who attended the Survive & Thrive course designed for survivors of interpersonal trauma who meets the inclusion criteria will be invited to take part in a semi-structured interview. This interview will explore their experience of this psychoeducational course.
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Each participant will attend a 30-45 minute semi-structured interview conducted by the CI

SUMMARY:
The study is aimed to explore female patients' experience of the Survive & Thrive course that has been designed for survivors of interpersonal trauma (e.g. childhood sexual abuse, domestic abuse, rape, physical abuse, neglect, harassment, stalking and similar). The course aims to help attendees develop an understanding of the normal range of reactions to trauma and introduce new ways of coping. It is a 10 week course that is structured to utilise cognitive behavioural skills training while delivering psychoeducation on how a history of victimisation can impacts on the survivors life. Female adult participants who attended the Survive & Thrive course will be invited to take part in a 30-45 minutes semi-structured interview exploring their experience of the course. The aim is to interview 12 participants; those individuals attended 6 or more sessions. Access to some demographic information will be gained through the Survive & Thrive team to gain additional insight to the participant's course experience. The rationale for this study is to evaluate the effectiveness of the Survive & Thrive course as a treatment option within the Stepped Care Approach for survivors of interpersonal trauma. There is an increasing number of individuals being exposed to traumatic life events. Most research has concentrated on the individual psychological input for patients with trauma history. Courtois and Ford (2009) argued that at a service level, group therapy is more efficient than individual as it can be offered more broadly. There is however limited research on the effectiveness of manualised approaches for the mental health and behavioural problems. Research shows that safety and stabilisation in trauma survivors can be achieved through psychoeducational approaches which emphasise present-time, coping strategies/skills, elimination of self-harming behaviour, control over acute symptoms, and increased self-care (Lubin & Johnson, 1997). Findings from this study will be published.

DETAILED DESCRIPTION:
Design The proposed research is a qualitative study using a purposive sample (participants have a position of shared experience), consisting of semi-structured interviews and some demographic information will be collected from the Survive & Thrive database.

Procedures All the procedures planned for this research project have been considered in detail to ensure that they follow the highest standards in the BPS (2009) ethical guidelines and the Health & Care Professions Council (HCPC, 2012) standards of proficiency. Initially, the Survive & Thrive database will be screened by the Survive & Thrive course team for female patients who have attended any 6 or more sessions out of the 10. These sessions are not required to be consecutive. Each session co-facilitators record attendance that is then stored on the Survive & Thrive SMF. They will be sent a letter informing them of this study along with a participants' information sheet and a reply slip passing on their note of interest to be contacted by the CI about the study (please see attached documents). This letter will be sent by the Survive & Thrive team leader who was in prior contact with the patients and her name has been on prior correspondence with them. It will provide them with space to specify their preferred method of contact. A pre-paid envelope addressed to the CI will be provided. Once reply slip is received, I will contact them to offer further information about the study and arrange to meet with them to complete the consent form and to conduct the semi-structured interview. Please see attached forms that will be sent out to potential participants.

Additionally, co-facilitators will inform current patients about this study at the beginning of week 6 of the Survive & Thrive course and hand out the information sheet and reply slip. At the beginning of week 7, co-facilitators will ask patients to pass on the reply slip if they would like to be contacted by the CI to find out more about the study. The co-facilitators will be provided with an additional form that they will complete along with the attendance sheet (please see attached). This form will enable monitoring of who was informed of the study and who has agreed to be contacted in relation to it. All of the entries in this form will be initialled and dated by the Survive & Thrive co-facilitators. The CI will not have access to these forms and will only be provided with information & contact numbers for individuals who have shown interest in the study and agreed to be contacted in relation to it. When the CI contacts potential participants (upon receiving a reply slip) who have shown interest, it will be specified that the interview will be arranged after the 10th week of the course (once the course is completed). The potential participants had to attend during this time any 6 sessions or more of the 10 (not required to be consecutive).

If they agree to be contacted regarding this study, the CI will then contact them. The CI will provide them with additional information regarding the study that is detailed in the participant information sheet. Participants will be assured that all data is stored securely and confidentially. The demographic data will be given a code along with the interview transcript to match the two data sets.

Once the participants agree to take part, arrangements to meet at one of the clinical rooms will be made. At this point they will confirm their consent to participate in the study by signing the consent form. After they sign the consent form they will take part in the semi-structured interview. Lastly, the participants will take part in a brief off-tape discussion regarding their experience of the interview and thanked for their participation. A list of contact recommendations of who to contact if participants became distressed or would like further support/opportunity to speak about the topics discussed during the interview will be provided to them at the end of the interview.

Material Semi-structured interviews will be conducted. The choice of questions considered how best to reflect the chosen data analysis in IPA that is entirely concerned with understanding individuals' experiences, feelings, and meaning-making. Thus, the selected questions are concentrated on emotions, values, and priorities.

Methods of analysis The proposed method of analysis for this research project is Interpretative Phenomenological Analysis (IPA), a method that has particular resonance for psychologists within qualitative research. It offers an established, systematic, and phenomenologically-focused approach to the interpretation of first-person accounts. It is a meaning-focused qualitative method that is committed to the understanding of the first-person perspective of their experience from the third-person position through inter-subjective inquiry and analysis.

Analysis of the data gathered will begin with transcribing the twelve 30-45minutes semi-structured interviews (by the Service admin staff who types up clinical letters). A decision to use the NHS admin staff for transcribing of the interviews was made due to a time restriction on this research and to ensure for confidentiality of the data. This will provide some time security as well as ensuring that the transcript will be to the highest standard. Once the interviews are transcribed, the audio recording will be deleted. I will then start familiarising myself with the transcriptions. This will be followed by a cyclical process of synthesis and analysis which will involve the reading and re-reading of the transcripts followed by exploratory manual coding (no use of software) of anything of interest within the transcript that allows me to identify the specific ways each participant talks about, thinks about and understands their experience. This step is followed by identifying the emerging themes throughout the transcripts. Once these are identified I will draw a map of the emerging themes to provide a structure for writing up the information and clustering all the themes that are repeated.

Once this is completed I will go back over the gained information and start making sense of the data by connecting patterns and making connections between recurrent themes by looking at, for example, how these recurrent themes inter-relate. I will attempt to conceptualise the connections and patterns and use this to organise the data, and draw relationships between them. The production of a summary table is seen as a beneficial next step to gain a clear and systematic overview of thematic clusters, together with keywords and the locations of relevant quotations. Afterwards the interpretative part of the IPA, that has recently been divided into two distinct levels, begins. The first level is a more descriptive, empathic level, aiming to enter the participants' world, while the second level is seen as more critically interrogative of the participants' views, in order to gain further insight into their nature, meaning and origins. I will aim to draw predominantly on the first level of interpretation of the data as the second has received some ethical criticism around the imposition of meaning upon data.

Once writing up the findings some example quotations will be used to represent recurrent themes, to offer readers an insight into the survivors of interpersonal trauma who attended Survive & Thrive course thinking patterns. Excel (Microsoft office) program will then be used to conduct how many themes occur across how many participants.

ELIGIBILITY:
Inclusion Criteria:

* meet Survive & Thrive course criteria
* adults between the ages of 18 - 65 years
* able to consent
* history of interpersonal trauma (childhood sexual abuse, domestic abuse, rape, physical abuse, neglect, harassment, stalking and similar).
* attended 6 or more sessions of the course

Exclusion Criteria:

- individuals in cohorts facilitated by the chief investigator

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Bartoskova, Dr, Principal Investigator — NHS Tayside - Dundee Adult Psychological Therapies Service
Locations (1):
- Dundee Adult Psychological Therapies Service, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not applicable. Summary of anonymised quotes from the research study will be published

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Semi-structured Interview
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Semi-structured Interview
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 37.3 [19 to 62]
Sex: Female, Male [Count of Participants; unit: Participants] — Female participants only
  Participants
    Female | 13
    Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Participants Experience of the Survive & Thrive Course - Themes
Description: Total of 13 participants attended 30 minutes semi-structured interview which explored their experience of the Survive & Thrive course. The transcribed interviews were analysed using Interpretative Phenomenological Analysis (IPA). Superordinate themes captured by the interviews followed by respective sub-themes were:
  1. Sense of connectedness, Sub-themes: I am not alone; Shared understanding; Safe environment/space
  2. Journey towards recovery, Sub-themes: It gets harder before it gets better; Life changing experience; Sense of empowerment; Long way to go
  3. Facing the facts & triggers, Sub-themes: Facing denial & triggers; Eye opening moments; Acceptance and greater understanding
  4. Initial apprehension, Sub-themes: Sense of helplessness; Readiness for change; Fear of the unknown
  5. Sense of being let down, Sub-themes: Challenging personalities; Repetitiveness of questionnaires; Need for additional support
  The number of participants that fell into each theme are reported below.
Time Frame: 30-45 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Semi-structured Interview
Number analyzed (Participants) | 13
Participants
  Sense of connectedness | 12
  Journey towards recovery | 12
  Facing the facts & triggers | 13
  Initial apprehension | 13
  Sense of being let down | 4

ADVERSE EVENTS:
Time Frame: The study did not collect information on adverse event data.
Description: The study did not collect information on adverse event data.
Arm/Group | Semi-structured Interview
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT03649867/Prot_SAP_000.pdf